CLINICAL TRIAL: NCT06184334
Title: Assessment of Efficacy of Mirabegron, Solifenacin, Tadalafil 5mg and Combination Therapy in Female Patients With Overactive Bladder: A Double Blinded Prospective Randomized Placebo -Controlled Trial
Brief Title: Management of OAB in Female Patients .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsayed Abdelhalim Elsayed (Other)
Responsible Party: Sponsor-Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer, urology department, Kafrelsheikh university, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OAB
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A : patients will receive mirabegron (Active Comparator): patients will receive mirabegron
  Interventions: Drug: Mirabegron
- Group B: patients will receive tadalafil 5mg (Active Comparator): patients will receive tadalafil 5mg
  Interventions: Drug: Tadalafil 5mg
- Group C: patients will receive solfenacin (Active Comparator): patients will receive solfenacin
  Interventions: Drug: Solfenacin

INTERVENTIONS:
Drug: Solfenacin — pills taken once day
  Arms: Group C: patients will receive solfenacin
Drug: Mirabegron — pills taken once day
  Arms: Group A : patients will receive mirabegron
Drug: Tadalafil 5mg — pills taken once day
  Arms: Group B: patients will receive tadalafil 5mg

SUMMARY:
The objective of this study is to compare the effectiveness of mirabegron, solifenacin, tadalafil (5mg), and their combination in relieving symptoms of overactive bladder (OAB) in a double-blinded prospective randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 65 years of age with LUTs due to OAB

Exclusion Criteria:

* Severe cardiovascular disorders. \

  * Severe neurogenic dysfunction.
  * Drug administration which interfere with bladder function .
  * Abnormal bleeding profile.
  * A verified urinary tract infection as determined by urinalysis and/or urine culture during screening

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
overactive bladder symptoms score (OABSS) | three months
  OABSS is a symptom assessment questionnaire designed to quantify OAB symptoms into a single score The questionnaire consists of 4 questions on OAB symptoms with maximum scores ranging from 2 to 5: daytime frequency (2 points), night-time frequency (3 points), urgency (5 points), and UUI (5 points). The total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University hospital, Kafr ash Shaykh, Egypt